CLINICAL TRIAL: NCT03437447
Title: A Phase I, Open-label, Randomized, Three-period, Crossover, Partial Replicated, Reference-scaled, Single Center Trial to Assess the Bioequivalence of a Single Oral Dose of 1200 mg of the New Cisticid 600 mg Tablet Formulation Versus Comparator Biltricide in Healthy Male Volunteers
Brief Title: Praziquantel Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200585_0002
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Bioavailability; Bioequivalence; Praziquantel; Cysticide; Pharmacokinetics
MeSH Terms: interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Cisticid, Then Biltricide, Then Biltricide (Experimental): Cisticid (Test) in Treatment Period 1 followed by Biltricide (Reference) in Treatment Period 2 and Treatment Period 3. A washout period of 7 days will be maintained between 3 treatment periods.
  Interventions: Drug: Cisticid; Drug: Biltricide
- First Biltricide, Then Cisticid, Then Biltricide (Experimental): Biltricide (Reference) in Treatment Period 1 followed by Cisticid (Test) in Treatment Period 2 and then Biltricide (Reference) in Treatment Period 3. A washout period of 7 days will be maintained between 3 treatment periods.
  Interventions: Drug: Cisticid; Drug: Biltricide
- First Biltricide, Then Biltricide, Then Cisticid (Experimental): Biltricide (Reference) in Treatment Period 1 and Treatment Period 2 followed by Cisticid (Test) in Treatment Period 3. A washout period of 7 days will be maintained between 3 treatment periods.
  Interventions: Drug: Cisticid; Drug: Biltricide

INTERVENTIONS:
Drug: Cisticid — Participants received single oral dose of 1200 mg (two 600 mg tablets) Cisticid (Test) on Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2) or Day 15 (Treatment Period 3).
  Other Names: Praziquantel
Drug: Biltricide — Participants received 600 mg of Biltricide (Reference) tablet at a dose of 1200 mg on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
  Other Names: Praziquantel

SUMMARY:
The purpose of this trial is to assess the bioequivalence (BE) of new 600 milligram (mg) Cisticid tablet (Test) versus 600 mg Biltricide tablets (Reference) at a dose of 1200 mg in healthy male participants. Praziquantel (PZQ) is the active ingredient for Cisticid and Biltricide tablets.

ELIGIBILITY:
Inclusion Criteria:

* A male participant must agree to use and to have their female partners willing to use additional non-hormonal contraception (for example, condoms or occlusive cap with spermicide, non-hormonal intra-uterine device [IUD], previous sterilization of participant or his partner, being sexually inactive) from Day of randomization up to final end of treatment (EOT) visit
* Gave written informed consent prior to any trial related procedure
* Have a body weight (BW) of greater than (>) 55.0 kilogram (kg) to less than (<) 95 kg and a body mass index (BMI) between 18.0 and 27.0 kg/meter square (m^2)
* Able to communicate well with the Investigator, understanding the protocol requirements and restrictions, and willing to comply with the requirements of the entire trial
* Non-smoker (= 0 cigarettes, pipes, cigars or others) since at least three months
* Electrocardiogram recording (12-lead) without signs of clinically relevant pathology in particular heart-rate corrected [QTc] (Bazett) <450 milliseconds (ms)
* Vital signs should be in normal range (systolic blood pressure: 90 to 140 millimeters of mercury [mmHg]; diastolic blood pressure: 50 to 90 mmHg; pulse rate: 45 to 90 beats per minute [bpm]; oral body temperature between 35.0 degree centigrade [°C] to 37.5°C)
* All values for biochemistry, liver function test and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator. Hematocrit and hemoglobin must be above the lower limit; upper limit may range up to 15 percent (%). Remaining results, including white blood cells may range +/- 15%, if participant is asymptomatic
* Negative screen for alcohol and drugs of abuse (opiate class, barbiturates, cocaine and metabolites, amphetamines, cannabinoids, benzodiazepines and tricyclic antidepressants) at screening and on each admission
* Negative screen for Hepatitis B surface (HBs) antigens, Hepatitis C Virus (HCV) antibodies, Hepatitis A Virus (HAV) antibodies and Human Immunodeficiency Virus (HIV) 1 and 2 antibodies
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* History of surgery of the gastrointestinal (GI) tract, history of other GI tract diseases, or acute GI tract infections in the last 2 weeks, which could influence the gastrointestinal absorption and/or motility according to the Investigator's opinion
* Any clinically relevant abnormality in the safety laboratory parameters as judged by the Investigator
* Have positive results from serology examination for Hepatitis B surface (HBs) antigen, Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Allergy: ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the trial
* History or presence of drug abuse (opiate class, barbiturates, cocaine and its main metabolite, amphetamines, cannabinoids, benzodiazepines and tricyclic antidepressants) or alcohol abuse at screening and on each admission. Alcohol abuse is defined by the assessment of the Investigator
* Loss or donation of more than 400 milliliter (mL) of blood within 90 days prior to first Praziquantel (PZQ) administration
* Administration of any investigational product or use of any investigational device in any clinical study within 30 days prior to first PZQ administration. Participants who have used drugs that may affect the pharmacokinetics of PZQ from 14 days before dosing until the last pharmacokinetic (PK) sample, for example, phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, oral ketoconazole
* Consumption of substances known to be potent inhibitors or inducers of Cytochrome P450s (CYP P450s) such as grapefruit, orange, cranberry or juices of these fruits, herbal remedies or dietary supplements containing St. John's Wort, poppy seeds, cruciferic vegetables, in the two weeks before dosing until last PK sample
* Unlikely to comply with the protocol requirements, instructions and trial-related restrictions, for example, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial
* Non-acceptance or non-compliance with the study breakfast (for example, vegetarians, vegans and participants who follow special diets)
* Excessive consumption of beverages containing xanthine (>5 cups of coffee a day or equivalent) or inability to stop consuming caffeine from 48 hours prior to drug administration until discharge from the clinic
* Participant is the Investigator or any Sub-Investigator, research assistant, pharmacist, trial coordinator, other staff or relative thereof directly involved in the conduct of the trial
* Vulnerable participants (for example, persons kept in detention)
* Legal incapacity or limited legal capacity
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Clínica de Enfermedades Crónicas y de Procedimientos Especiales, Sociedad Civil (SC), México, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- First Cisticid, Then Biltricide, Then Biltricide: Participants received single oral dose of 1200 milligrams (mg) (two 600 mg tablets) Cisticid (Test) on Day 1 in Treatment Period 1 followed by single oral dose of 1200 mg (two 600 mg tablets) of Biltricide (Reference) on Day 8 in Treatment Period 2 and on Day 15 in Treatment Period 3. A washout period will be maintained between 3 treatment periods.
- First Biltricide, Then Cisticid, Then Biltricide: Participants received single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference) on Day 1 in Treatment Period 1 followed by single oral dose of 1200 mg (two 600 mg tablets) of Cisticid (Test) on Day 8 in Treatment Period 2 and then single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference) on Day 15 in Treatment Period 3. A washout period will be maintained between 3 treatment periods.
- First Biltricide, Then Biltricide, Then Cisticid: Participants received single oral dose of 1200 mg (two 600 mg tablets) Biltricide (Reference) on Day 1 in Treatment Period 1 and on Day 8 in Treatment Period 2 followed by single oral dose of 1200 mg (two 600 mg tablets) of Cisticid (Test) on Day 15 in Treatment Period 3. A washout period will be maintained between 3 treatment periods.
Period: Treatment Period 1
Arm/Group | First Cisticid, Then Biltricide, Then Biltricide | First Biltricide, Then Cisticid, Then Biltricide | First Biltricide, Then Biltricide, Then Cisticid
Started | 20 | 20 | 20
Completed | 20 | 20 | 19
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | First Cisticid, Then Biltricide, Then Biltricide | First Biltricide, Then Cisticid, Then Biltricide | First Biltricide, Then Biltricide, Then Cisticid
Started | 20 | 20 | 19
Completed | 20 | 20 | 19
Not Completed | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | First Cisticid, Then Biltricide, Then Biltricide | First Biltricide, Then Cisticid, Then Biltricide | First Biltricide, Then Biltricide, Then Cisticid
Started | 20 | 20 | 19
Completed | 20 | 20 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Cisticid, Then Biltricide, Then Biltricide | First Biltricide, Then Cisticid, Then Biltricide | First Biltricide, Then Biltricide, Then Cisticid | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All participants who were randomized into the study.
  Years | 27.80 (7.83) | 28.65 (7.46) | 27.20 (5.31) | 27.88 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants who were randomized into the study.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 20 | 20 | 20 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants who were randomized into the study.
  Participants
    Hispanic or Latino | 20 | 20 | 20 | 60
    Not Hispanic or Latino | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants who were randomized into the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 20 | 20 | 20 | 60
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of L-Praziquantel (L-PZQ)
Description: Area under the plasma concentration-time curve from 0 to the time of the last quantifiable concentration.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 8.0, 9.0, 10.0 and 12.0 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all participants who received all administrations of treatment and have PK parameters for AUC0-t and maximum observed plasma concentration (Cmax) in all periods and without any relevant protocol violations and factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter (h*ng/ml)
Groups:
- Cisticid: All participants who received single oral dose of 1200 mg (two 600 mg tablets) Cisticid (Test) on Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2) or Day 15 (Treatment Period 3).
- Biltricide First Administration: All participants who received 600 mg of Biltricide (Reference) tablet at a dose of 1200 mg on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
- Biltricide Second Administration: All participants who received 600 mg of Biltricide (Reference) tablet at a dose of 1200 mg on either Day 8 (Treatment Period 2) or Day 15 (Treatment Period 3).
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
Hour*nanogram per milliliter (h*ng/ml) | 441.53 (345.70) | 547.41 (384.82) | 460.25 (343.37)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of L-Praziquantel (L-PZQ)
Description: The maximum observed plasma concentration of L-Praziquantel (L-PZQ).
Time Frame: as for outcome 1
Population: PK analysis set included all participant who received all administrations of treatment and have PK parameters for AUC0-t and Cmax in all periods and without any relevant protocol violations and factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
ng/mL | 310.87 (249.02) | 426.42 (324.01) | 363.20 (333.50)

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Time of the maximum drug concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
hours
  L-PZQ | 2.5 [1.5 to 5.5] | 2 [1 to 3.5] | 2.5 [1 to 4.5]
  Rac-PZQ | 2.5 [1.5 to 5.5] | 2 [1 to 3.5] | 2.5 [1 to 4.5]

4. Secondary Outcome: Time Prior to the First Measurable (Non-zero) Concentration (Tlag) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Time prior to the first measurable (non-zero) concentration; calculated as last time point at which the concentration is less than (<) Lower Limit of Quantification (LLOQ) before the occurrence of the first quantifiable concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
hours
  L-PZQ | 1 [0.25 to 3] | 1 [0.25 to 2.5] | 1 [0.25 to 3.5]
  Rac-PZQ | 0.75 [0.00 to 2.00] | 0.75 [0.25 to 2.00] | 0.75 [0 to 2.5]

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: AUC0-inf is defined as the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: as for outcome 1
Population: PK analysis set: All participants who received all administrations of treatment & have PK parameters for AUC0-t & Cmax in all periods without any relevant protocol violations & factors likely to affect comparability of PK results. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure for specified category.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
h*ng/ml
  L-PZQ: number analyzed (Participants) | 58 | 58 | 57
  L-PZQ | 468.52 (352.29) | 584.23 (410.05) | 497.89 (348.81)
  Rac-PZQ | 2130.19 (1417.81) | 2509.42 (1624.33) | 2189.25 (1403.14)

6. Secondary Outcome: Extrapolated Area Under the Plasma Concentration Curve From Time Tlast to Infinity (AUCextra) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of AUC0-inf
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
Percentage of AUC0-inf
  L-PZQ: number analyzed (Participants) | 58 | 58 | 57
  L-PZQ | 5.36 (3.73) | 5.49 (6.47) | 5.74 (4.02)
  Rac-PZQ | 2.60 (1.73) | 2.84 (2.56) | 2.57 (1.56)

7. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
hours
  L-PZQ: number analyzed (Participants) | 58 | 58 | 57
  L-PZQ | 1.87 (1.12) | 2.59 (3.01) | 2.32 (1.65)
  Rac-PZQ | 2.19 (0.91) | 2.54 (1.73) | 2.18 (0.90)

8. Secondary Outcome: Terminal Elimination Rate Constant (Lambda Z) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Lambda Z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: PK analysis set included all participants who received all administrations of treatment and have PK parameters for AUC0-t and Cmax in all periods and without any relevant protocol violations and factors likely to affect the comparability of PK results.
Measure: Median (Full Range); unit: Per hour
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
Per hour
  L-PZQ | 0.452927 [0.103378 to 1.120808] | 0.383267 [0.032567 to 0.721124] | 0.370854 [0.073375 to 0.944209]
  Rac-PZQ | 0.365639 [0.135661 to 0.646499] | 0.331359 [0.060282 to 0.635357] | 0.370806 [0.125134 to 0.638226]

9. Secondary Outcome: Apparent Clearance (CL/f) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Milliliter per hour
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
Milliliter per hour
  L-PZQ: number analyzed (Participants) | 58 | 58 | 57
  L-PZQ | 749261.50 (744206.88) | 585260.42 (541013.95) | 673193.51 (531848.19)
  Rac-PZQ | 147268.6 (122977.13) | 128110.14 (122864.03) | 155851.99 (145104.37)

10. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vd/f) of L-Praziquantel (L-PZQ) and Racemate PZQ (Rac-PZQ)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vd/f after oral dose was influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
Milliliter
  L-PZQ: number analyzed (Participants) | 58 | 58 | 57
  L-PZQ | 1540237.10 (1069504.21) | 1660474.33 (1619772.26) | 1800582.47 (1385707.17)
  Rac-PZQ | 430368.23 (328721.73) | 385223.26 (279076.69) | 431494.33 (350782.53)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Racemate PZQ (Rac-PZQ)
Description: Area under the drug plasma concentration-time curve from time zero to the time last measurable concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
h*ng/ml | 2071.35 (1370.58) | 2421.73 (1518.94) | 2131.01 (1353.64)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Racemate PZQ (Rac-PZQ)
Description: The maximum observed plasma concentration of rac-Praziquantel (rac-PZQ).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 59 | 59 | 59
ng/mL | 1209.15 (803.20) | 1530.23 (944.12) | 1356.18 (1011.46)

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 29
Population: Safety Analysis Set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 60 | 60 | 60
Participants
  Participants with TEAEs | 2 | 5 | 6
  Participants with Serious TEAEs | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Number of participants with clinically significant abnormalities in laboratory parameters were reported. Laboratory investigation included hematology, biochemistry, urinalysis and coagulation.
Time Frame: Baseline up to Day 29
Population: Safety Analysis Set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 60 | 60 | 60
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs were reported. Vital signs included body temperature, systolic / diastolic blood pressure, and pulse rate.
Time Frame: Baseline up to Day 29
Population: Safety Analysis Set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 60 | 60 | 60
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with clinically significant abnormalities in 12-lead electrocardiogram (ECG) were reported. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position.
Time Frame: Baseline up to Day 29
Population: Safety Analysis Set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
Number analyzed (Participants) | 60 | 60 | 60
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29
Arm/Group | Cisticid | Biltricide First Administration | Biltricide Second Administration
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 2/60 | 5/60 | 6/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisticid (N=60) | Biltricide First Administration (N=60) | Biltricide Second Administration (N=60)
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1
Alanine Transaminase Increased (Investigations) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03437447/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03437447/SAP_001.pdf